CLINICAL TRIAL: NCT06709482
Title: Predicting Postoperative Delirium With Heart Rate Variability Obtained by Analgesia Nociception Index - A Prospective Clinical Pilot Study
Brief Title: Predicting Postoperative Delirium With Heart Rate Variability Obtained by Analgesia Nociception Index
Acronym: DANI
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: EK Nr: 1061/2024
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-11

CONDITIONS: POSTOPERATIVE DELIRIUM AND POSTOPERATIVE COGNITIVE DECLINE; Heart Rate Variability; Biomarkers
Keywords: postoperative delirium; inflammation; heart rate variability
MeSH Terms: conditions — Emergence Delirium; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this pilot study is to establish a correlation between perioperative heart rate variability (HRV) as an expression of the shift in the balance of the autonomic nervous system and the occurrence of postoperative inflammation and delirium. The main question it aims to answer is: Do patient with increased sympathetic nervous system activity develop postoperative delirium (POD) more often than patients with increased parasympathetic tone?

DETAILED DESCRIPTION:
Cholinergic failure is a function of human aging that is associated with neurocognitive disorders, including delirium and the most common dementia, Alzheimer's disease. Although the exact mechanisms involved in the development of delirium are still poorly understood, an abnormal stress response and neurotransmitter imbalance, especially acetylcholine, as well as age-related changes in the decline of the parasympathetic system, increased levels of (neuro)inflammation, and reduced resilience of the human brain are considered crucial elements in the pathophysiology of delirium. Therefore, elderly patients undergoing surgery are at increased risk of developing postoperative delirium (POD) and postoperative cognitive dysfunction (POCD). Several risk factors for the development of POD are currently discussed, including older age, neurocognitive impairment, frailty, comorbidity, neurological or psychiatric disease. The available scientific evidence, mostly from animal studies but also from a few human studies, emphasizes that the induction of neuroinflammation in the central nervous system is triggered by surgical trauma. The vagal nerve coordinates most physiological functions, including the cardiovascular and immune systems. Peripheral cytokines can stimulate the afferent vagal nerve and stimulate the reciprocal response of the hypothalamic-pituitary-adrenal axis and anti-inflammatory vagal activities (via α7nACHR on macrophages in the spleen, which inhibits cytokine production). This mechanism has significant clinical implications because electrical stimulation of the vagal nerve can control inflammation and organ injury in infectious and inflammatory diseases. Vagal nerve stimulation prevents organ injury and systemic inflammation by inhibiting cytokine production in the spleen.

Recent physiological and anatomical studies suggest that inflammation is regulated by neuroimmune multi-synaptic interactions between the vagal and splanchnic nerves to modulate the spleen. In contrast to the role of the parasympathetic vagal nerve, the innervation of the spleen by the splenic sympathetic nerve has been well documented by a number of neuroanatomical studies in various species, including rodents, cats, and humans. Several clinical studies are underway showing that electrical vagal stimulation is a promising approach for the treatment of chronic inflammatory diseases. Vagal nerve stimulation reduced blood markers of inflammation such as C-reactive protein and fecal calprotectin, improved mood, clinical symptoms of rheumatoid arthritis, and significantly reduced serum levels of inflammatory cytokines. Patients with delirium have an abnormal autonomic nervous system response as assessed by ECG recordings and the head-up tilt test. These patients show parasympathetic dysfunction in delirious patients (in the ICU and postoperatively). For example, there is a correlation between preoperative heart rate variability and the development of POD in patients aged 65 years or older undergoing planned open-heart surgery, with the high-frequency components of the ECG, considered to be parasympathetic nerve activity, being reduced in delirious patients. Thus, the onset of POD may be associated with the preoperative functional decline of autonomic nerves, especially parasympathetic nerves.

THE ANALGESIA NOCICEPTION INDEX The Analgesia Nociception Index (ANI™, Mdoloris Medical Systems, Loos, France) is a relatively new technology designed to assess intraoperative pain during general anesthesia. The system provides measurement of parasympathetic tone and evaluation of the sympathetic-parasympathetic balance during surgery derived from the ECG. Because surgical stress affects the sympathetic-parasympathetic balance, which can be detected by a change in heart rate variability (HRV). The influence of surgical stress on HRV and a shift of the autonomic nervous system towards sympathetic activity has been shown in several studies.

The (neuro)inflammatory hypothesis of delirium is supported by biomarker studies showing increased levels of cytokines and neuroaxonal damage markers in patients with POD. However, the interplay between surgical stress and inflammation leading to parasympathetic-sympathetic imbalance and cholinergic dysfunction resulting in neuroinflammation remains to be characterized in depth. To our knowledge, this will be the first study to correlate the autonomic nervous system by ANI™ monitoring with multiple serum markers involved in neuronal damage, neuroinflammation and stress response.

The purpose of the following pilot study is to evaluate heart rate variability (HRV), indicative of sympathetic-parasympathetic balance, using ANI™ monitoring before, during, and after anesthesia and its relationship to POD in patients undergoing moderate to high risk orthopedic or trauma surgery.

PRIMARY OBJECTIVES:

1. Characterize the sympathetic-parasympathetic balance by ANI™ monitoring (pre-, during and post-operative) in elective orthopedic surgery patients and its relationship to the incidence and severity of POD and POCD, AND
2. To evaluate cognition and cognitive decline 90 days after surgery in elective orthopedic surgery patients with and without POD, AND
3. To evaluate serum concentrations of (neuro-)inflammatory and neurodegenerative markers, including interleukins and S-100B, NSE, NfL, among other potential biomarkers, together with coagulation factor concentrations and hemostasis parameters in elective orthopedic surgery patients with and without POD/POCD.
4. Correlate serum-derived markers with the incidence and severity of POD/POCD and ANI(TM) monitoring and determine if ANI(TM) monitoring can indicate perioperative inflammation and predict POD/POCD, 5.) To evaluate preoperatively assessed personality traits, frailty, depression, and anxiety in elective orthopedic surgery patients with and without POD/POCD to determine whether their predictive value with respect to POD/POCD.

6.) Correlation of gender differences in HRV and neuroinflammation will be assessed at all study stages and subgroup analysis will be performed. Results will be published according to SAGER guidelines.

PATIENTS´ DEMOGRAPHICS AND MEDICAL HISTORY:

Eligible patients will be identified and after obtaining informed consent, basic demographic data (age, sex, education, body mass index, sex, ethnicity, American Society of Anesthesiology physical status) as well as social history including tobacco use, comorbidities, long-term medications, and type of surgery will be recorded.

COGNITION:

One hundred and fifty (75 participants aged 50-75 years and 75 patients >75 years) individuals will be enrolled in this pilot study. Patients will undergo a detailed neurocognitive assessment by neuropsychologists using a battery of tests including CERAD (Consortium to Establish a Registry for Alzheimer's Disease); MoCA (Montreal Cognitive Assessment); CAM/CAM-ICU/3D-CAM (various forms of the Confusion Assessment Method); DOS (Delirium Observation Scale); BPI (Behavioral Pain Scale); CPOT (Critical Pain Observation Tool); GDS (Geriatric Depression Scale); BFI-10 (Big Five Inventory-10); DRSR-98 (Delirium Rating Scale -Revised-98); NRS (Numerical Rating Scale); EQ-5D-5L (Health Questionnaire).

QUESTIONNAIRES AND RATING SCALES:

The following scores and assessments will be performed by a trained person:

* The Barthel Index
* The Numeric Rating Scale (NRS)
* The Behavioral Pain Inventory (BPI)
* The Critical Care Pain Observation Tool (CPOT)
* The Big Five Inventory (BFI-10;)
* The Clinical Frailty Scale (CFS)
* Richmond Agitation Sedation Scale (RASS)
* Confusion Assessment Method (CAM/CAM-ICU)
* 3D CAM
* DOS
* Depression, Anxiety and Stress Scale (DASS)
* Geriatric Depression Scale Quality of life is assessed using
* the EQ-5D-5L

ANI™ MONITORING:

Baseline ANI™ monitoring will be administered the day before surgery and recorded for at least 5 minutes for all study participants.

DIAGNOSTIC WORKUP AND BLOOD SAMPLES:

In addition to blood samples for routine diagnostic workup, inflammatory markers i as well as biomarkers of neurogeneration/neuroinflammation and markers of blood-brain barrier disruption (neuron-specific enolase (NSE), S100B) will be measured.

INTRAOPERATIVE MANAGEMENT:

Routine intraoperative and postoperative anesthesia-specific data will be extracted from our electronic anesthesia records. Intraoperative monitoring of depth of anesthesia will be performed using the Bispectral Index (Bispectral Index™, Medtronic, Minneapolis, United States of America) and blinded ANI™ Monitoring.

POSTOPERATIVE SCREENING:

After surgery, patients will be screened for POD twice daily (morning between 5:00 am and 10:00 am and evening between 5:00 pm and 10:00 pm), as well as any time patients show a change in mental status. Patient alertness and activity will be characterized by the RASS scale.

Patients with intubated POD will be assessed by RASS and CAM-ICU. All other patients, POD will be evaluated by 3D-CAM/CAM and the DOS. In addition, the patient's chart will be reviewed for any symptoms that can be attributed to the POD and the CHART-DEL. The duration of POD and any interfering medications will be documented. The severity of POD is assessed using the 3DCAM and CAM-S. The subtype of POD will be assessed according to the patient's RASS score (RASS score of -4 or -5 will not be considered for delirium screening, hyperactive POD corresponds to a positive delirium screening and a RASS score > 0, hypoactive delirium will be considered if the RASS score is <1). Patients are considered delirious if they have a RASS greater than or equal to -3 and a positive CAM-ICU result. Subsyndromal POD will be assigned if the Confusion Assessment Method (CAM) or CAM-ICU score is positive on 1 or 2 items out of 4. Postoperative pain will be assessed using the Numerical Rating Scale (NRS) at the same time as delirium screening and medication will be recorded.

FOLLOW-UP:

Ninety days after surgery, patients will be invited for follow-up. All patients will be assessed using the MoCA, EQ-5D-5L questionnaire, DASS, GDS, CSF, Barthel Index and pain assessment. All subjects will undergo a structured neurocognitive assessment at the Department of Neurology, Innsbruck.

One year after surgery, patients will be contacted by telephone to obtain their Barthel Index and EQ-5D-5L.

STATISTICAL ANALYSIS:

SPSS will be used for statistical analysis. No sample size calculation was performed due to the exploratory nature of this pilot study and the unknown effects of ANI™ monitoring. An interim analysis will be performed after 75 patients have been enrolled and the study may be terminated at that time. Descriptive statistics will be used to characterize the study population and groups. Depending on the distribution of the data (parametric versus non-parametric), either the confidence interval and range or the mean and standard deviation will be calculated. Frequencies and odds ratios are calculated using crosstabs and chi-squared tests. Subgroup analyses will be performed with respect to preoperative cognitive function, comorbidities, and medications. Group differences comparing two groups will be assessed using Student t test or Mann-Whitney U test, as appropriate. For comparisons of more than two groups, one-way ANOVA or Kruskal-Wallis test with post hoc Bonferroni test will be used. Receiver operating curve analyses will be performed for the candidate serum markers. The predictive value of candidate serum proteins, ANI™, frailty, personality traits for the occurrence of delirium and postoperative cognition will be assessed by logistic regression analyses. Pearson or Spearman rank test will be calculated to assess correlations. The significance level will be set at p<0.05.

RISK ASSESSMENT:

A total of 140 ml of blood will be collected throughout the study period from baseline to 90 days after surgery. There is no additional health risk to participants from the use of ANI™ monitoring, clinical questionnaires, and rating scales. If dementia is diagnosed, patients will be offered the opportunity to present at the Memory Outpatient Clinic.

ELIGIBILITY:
Inclusion Criteria:

1. > 50 years of age
2. Scheduled for elective moderate to major risk traumatology or orthopedic surgery (excluding spine surgery) and anticipated duration of general anaesthesia ≥ 60 minutes.

Exclusion Criteria:

1. Delirium before surgery.
2. Patients with emergency surgery
3. Contraindication to general anesthesia
4. ASA ≥ 4.
5. Terminal disease.
6. h/o documented dementia, MoCA Score <18
7. h/o atrial fibrillation
8. h/o Parkinson´s disease / Multiple system atrophy / Pure autonomic failure
9. h/o autonomic dysfunction (neurogenic autonomic dysfunction)
10. h/o stroke/intracerebral hemorrhage
11. Cerebral neoplasia
12. h/o chronic central nervous disorder (e.g. multiple sclerosis)
13. Major Depression
14. Language, vision, or hearing impairments that may compromise delirium or cognitive assessments.
15. h/o malignant hyperthermia
16. h/o structural muscle disease
17. h/o substance abuse
18. h/o polyneuropathy
19. h/o psychiatric disease
20. h/o or current substance use disorder (DSM V)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients > 50 years undergoing surgery lasting at least 60 min
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive function at 90 days after surgery | 90 days
  Structured neurocognitive assessment using the test battery.

SECONDARY OUTCOMES:
HRV and postoperative delirium | 5 days
  Comparison of heart rate variability before, during and after anaesthesia in patients with and without POCD.

OTHER OUTCOMES:
neuro-degenerative/neuro-inflammation markers inflammatory | 90 days
  Correlation of the concentration of the biomarkers S-100B (µg/L), NSE (µg/L), NfL (pg/mL), CRP (mg/L) PCT (mg/L), IL-6 (pg/mL), TNF-alpha (ng/mL), in patients with and without POD/POCD

CONTACTS AND LOCATIONS:
Overall Officials: Christine Eckhardt, MD, PhD, Principal Investigator — Medical University Innsbruck

IPD SHARING:
Plan to Share IPD: Undecided